CLINICAL TRIAL: NCT00081341
Title: Cognition, Steroids, and Imaging in Cushings Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: 51337DK (completed)
Record Dates: First submitted 2004-04-08; First posted 2004-04-12 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Cushing Syndrome
MeSH Terms: conditions — Cushing Syndrome

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study investigates the effects of the glucocorticoid hormone cortisol on brain structure and function. Patients with Cushing's disease are studied before and after treatment. Brain imaging and neuropsychologic tests are used to study changes in the hippocampus and thinking and learning functions as well as mood during the period of elevated cortisol. At several intervals after treatment, these are reexamined to study the degree of reversibility of the abnormalities. The contribution of cortisol as well as testosterone and estrogen to dysfunction and recovery is studied. Since elevated cortisol and dysregulation of its secretory system occurs in a significant proportion of the aged and in Alzheimers Disease and Major Depressive Disorder, these studies will help advance knowledge of the role of cortisol in these conditions.

ELIGIBILITY:
Inclusion criteria:

* patients with suspected Cushing's syndrome with clinical findings suggestive of Cushing's syndrome and positive screening tests (urinary free cortisol and low dose overnight dexamethasone suppression test).

Exclusion criteria: none

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- General Clinical Research Center, University of Michigan Health System, Ann Arbor, Michigan, United States